CLINICAL TRIAL: NCT02566525
Title: CytoSorb Reduction of Free Hemoglobin During Cardiac Surgery
Acronym: REFRESH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CytoSorbents, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-001
Record Dates: First submitted 2015-09-28; First posted 2015-10-02 (Estimated); Results first posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-07

CONDITIONS: Elective Cardiac Surgery
Keywords: CytoSorb device; Plasma free hemoglobin; inflammation; extracorporeal bypass
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CytoSorb Device (Experimental): Standard of care plus treatment with CytSorb device installed on the CPB machine
  Interventions: Device: CytoSorb
- Control (No Intervention): Standard of care

INTERVENTIONS:
Device: CytoSorb — Cytosorb device use during cardiopulmonary bypass
  Arms: CytoSorb Device

SUMMARY:
Prospective, multi-center, randomized, feasibility clinical study. Subjects will be randomized in a 1:1 ratio to either standard of care (SOC) alone or standard of care and treatment with the CytoSorb® device.

ELIGIBILITY:
Inclusion Criteria:

* Elective, cardiac surgery requiring cardiopulmonary bypass with anticipated duration of >180 minutes

Exclusion Criteria:

* Platelet count < 20,000/ uL
* Body mass index <18
* Pregnant women
* Life expectancy of <14 days
* End stage organ disease
* Active infection
* Undergoing cardiac transplant or ventricular assist device explant, isolated primary coronary artery bypass grafting (CABG) or single valve procedure
* Contraindication to anticoagulation with heparin
* Declined informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Sisk, MSc Pharm, Study Director — CytSorbents
Locations (8):
- United States (8):
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Baystate Medical, Springfield, Massachusetts
  - Cooper University Hospital, Camden, New Jersey
  - Columbia University, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Heymann M, Schorer R, Putzu A. The Effect of CytoSorb on Inflammatory Markers in Critically Ill Patients: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Crit Care Med. 2023 Dec 1;51(12):1659-1673. doi: 10.1097/CCM.0000000000006007. Epub 2023 Aug 21. PMID 37607074

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In; 8 December, 2015 Last Patient in: 19 August 2016
  Mostly university hospitals; all sites had robust cardiac surgery programs
Pre-assignment Details: Potential patients had to have a planned 3+ hour bypass time. Isolated coronary bypass graft or single valve procedures were excluded. Cases included were aortic reconstructions, valve repairs, valve replacements and combinations thereof, and permitted combination with coronary bypass graft. Emergency and endocarditis patients were excluded. 52 patients enrolled in the study, of which 6 withdrew from the study.
Groups:
- CytoSorb Device: Standard of care cardiac surgery with CPB plus treatment with CytSorb device installed on the CPB machine
  CytoSorb: Cytosorb device use during cardiopulmonary bypass
- Control: Standard of care, cardiac surgery patients, cardiac bypass with no CytoSorb device
Period: Overall Study
Arm/Group | CytoSorb Device | Control
Started | 23 (FPI - CytoSorb Patient 15 Jan 2016) | 23 (FPI - Control Patient 8 Dec 2015)
Completed | 20 (LPI - CytoSorb Patient 19 Aug 2016) | 18 (LPI - Control 16 Aug 2016)
Not Completed | 3 | 5
Not completed — Protocol Violation | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CytoSorb Device | Control | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.09 (7.91) | 61.09 (16.77) | 63.59 (13.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 13 | 18 | 31
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Serious Device Related Adverse Events
Description: The primary safety endpoint of this trial was to determine the product safety profile through the assessment of serious device related AEs through discharge from the ICU.
Time Frame: From time of enrollment through ICU discharge (e.g. ICU stay of approximately 4 days)
Population: All patients who had at least on Adverse Event
Measure: Number; unit: participants
Arm/Group | CytoSorb Device | Control
Number analyzed (Participants) | 23 | 23
participants
  Participants with at least one device related AE | 2 | 0
  Participants with at least one SAE | 16 | 11

2. Secondary Outcome: Time in the ICU
Description: Days in ICU, Post Surgery
Time Frame: From the end of cardiopulmonary bypass procedure through ICU discharge (e.g. ICU stay of approximately 4 days)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | CytoSorb Device | Control
Number analyzed (Participants) | 23 | 23
Days | 4.34 (3.34) | 6.82 (12.74)

3. Secondary Outcome: 30 Day All Cause Mortality
Description: Mortality within 30 Days of Surgery
Time Frame: From time of enrollment through 30 days post procedure
Population: All patients who were randomized to trial and had a surgical procedure
Measure: Number; unit: participants
Arm/Group | CytoSorb Device | Control
Number analyzed (Participants) | 23 | 23
participants | 2 | 1

4. Secondary Outcome: Adverse Event Rates
Description: Total number of Serious Adverse Events
Time Frame: through 30 days
Population: Total number of Serious Adverse Events
Measure: Number; unit: SAE
Arm/Group | CytoSorb Device | Control
Number analyzed (Participants) | 23 | 23
SAE | 44 | 43

5. Other Pre Specified Outcome: Change in Complement Factor C3a - 2 Hours Post Start of CPB
Description: Change in complement factor C3a - Sampling at 2 hours post start of CPB
Time Frame: 2 hours post start of cardiac bypass
Population: Patients with evaluable C3a laboratories
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | CytoSorb Device | Control
Number analyzed (Participants) | 20 | 21
ng/ml | 1146.75 (383) | 3116.24 (4008)

6. Other Pre Specified Outcome: Change in Complement Factor C3a - 3 Hours Post Start of CPB
Description: Change in complement factor C3a - Sampling at 3 hours post start of CPB
Time Frame: 3 hours post start of CPB
Population: Patients with evaluable C3a laboratory values at 3 hours post start of CPB
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | CytoSorb Device | Control
Number analyzed (Participants) | 15 | 10
ng/ml | 2491.1 (1339) | 1234.67 (424)

7. Other Pre Specified Outcome: Change in Complement Factor C5a - 2 Hours Post Start of CPB
Description: Change in complement factor C5a - Sampling at 2 hours post start of CPB, change from baseline
Time Frame: 2 hours post start of cardiac bypass
Population: Patients with evaluable C5a laboratories
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | CytoSorb Device | Control
Number analyzed (Participants) | 20 | 21
ng/ml | -7.29 (11.9) | 0.18 (3.98)

ADVERSE EVENTS:
Time Frame: Adverse events were reported for the 30 day period following Cardiac Surgery
Arm/Group | CytoSorb Device | Control
All-Cause Mortality (participants affected / at risk) | 2/23 | 1/23
Serious Adverse Events (participants affected / at risk) | 16/23 | 11/23
Other Adverse Events (participants affected / at risk) | 23/23 | 21/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CytoSorb Device (N=23) | Control (N=23)
Atrial Fibrilation (Cardiac disorders) | 2 | 2
Atrial flutter (Cardiac disorders) | 2 | 2
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 11
Right ventricular dysfunction (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac perforation (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Myocardial stunning (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Acute Lung Injury (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CytoSorb Device (N=23) | Control (N=23)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Atrial Fibrilation (Cardiac disorders) | 8 | 7
Atrioventricular block first degree (Cardiac disorders) | 1 | 2
Fluid overload (Metabolism and nutrition disorders) | 5 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3
Hypernatremia (Metabolism and nutrition disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 7
Leukocytosis (Blood and lymphatic system disorders) | 2 | 4
Coagulopathy (Blood and lymphatic system disorders) | 4 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Atalectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypotension (Vascular disorders) | 4 | 2
Haemorrhage (Vascular disorders) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 2
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute kidney injury (Renal and urinary disorders) | 5 | 5
Blood creatinine increased (Investigations) | 2 | 0
Tranaminases increased (Investigations) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 2
Ileus (Gastrointestinal disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No